CLINICAL TRIAL: NCT03324087
Title: A Multi-Center Prospective Study of Evaluating Health Related Quality of Life in Adult With Immune Thrombocytopenia in China Using Real-world Data
Brief Title: Evaluation of HRQoL in Adult With Immune Thrombocytopenia in China
Acronym: HRQoL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Qilu Hospital of Shandong University (Qingdao) (Other); Jining Medical University (Other); Liaocheng People's Hospital (Other); Yantai Yuhuangding Hospital (Other); Binzhou Medical University (Other); Weifang People's Hospital (Other); Linyi People's Hospital (Other); Shengli Oilfield Hospital (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Other Study IDs: ITP-HRQoL
Record Dates: First submitted 2017-08-21; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Immune Thrombocytopenia
Keywords: HRQoL; Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with ITP: The investigators are undertaking a multi-center, prospective trail of 1000 adult ITP patients and use SF-36 and ITP-PAQ questionnaires to assess the HRQoL in patients with ITP in the real world, and analyze the influencing factors of HRQoL so as to provide a sufficient basis for clinical decision making.
  Interventions: Diagnostic Test: HRQoL

INTERVENTIONS:
Diagnostic Test: HRQoL — use SF-36 and ITP-PAQ questionnaires to assess the HRQoL in patients with ITP in the real world, and analyze the influencing factors of HRQoL so as to provide a sufficient basis for clinical decision making.

SUMMARY:
Immune thrombocytopenia (ITP) is a heterogeneous disorder with variable clinical symptomsHealth related quality of life (HRQoL) could be considered in ITP, as in numerous chronic diseases, as a method to provide information about the effects of medical interventions. Symptoms of ITP, such as spontaneous bruising, menorrhagia, mucosal bleeding and prolonged bleeding with injury, may significantly affect HRQoL in ITP subjects. Treatments for chronic ITP can also be associated with substantial side effects. Restoring and/or maintaining quality of life should be an important goal of treatment. We conducted a real-world multicenter study using SF-36 and ITP-PAQ questionnaires to assess the HRQoL in patients with ITP in the real world, and analyze the influencing factors of HRQoL so as to provide a sufficient basis for clinical decision making.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an autoimmune thrombocytopenic syndrome characterized by decreased platelet count and an increased risk of bleeding.The pathogenesis of ITP has been considered as autoantibody-mediated and cell-mediated platelet over-destruction. The estimated prevalence for ITP in the China is 5-10/100,000. Adult women are disproportionately affected by the disorder, with a female to male ratio of nearly two to one. The disorder rarely remits spontaneously in adult subjects. The mortality rate is relatively low (< 1%) in adults less than 65 years of age. Morbidity increases above age 65, primarily as a result of an increase in age-related major bleeding events.

The decision to treat and the type of treatment are controversial, since among the different medications available, none has proven its superiority regarding reduction in bleeding complications or transition to chronic ITP. Furthermore, profound thrombocytopenia, the risk of intracranial bleeding, and the appearance of bruises may seriously influence lifestyle, school functioning and physical activities and frequently result in anxiety in children and adults. Therefore, since the benefit-risk ratio of current medications is unclear and as the psychological and the physical burden of the disease is highly variable, it appears necessary to develop new tools to better understand the exact impact of the disease on daily life. Although treatment decision making depends essentially on the physician's experience, it seems of interest to include in this reflection a measurement of quality of life. In this context, evaluation of health related quality of life (HRQoL) could be considered in ITP, as in numerous chronic diseases, as a method to provide information about the effects of medical interventions.

Symptoms of ITP, such as spontaneous bruising, menorrhagia, mucosal bleeding and prolonged bleeding with injury, may significantly affect HRQoL in ITP subjects. Treatments for chronic ITP can also be associated with substantial side effects. In addition, subjects who are resistant to current therapies are likely to experience an even greater decrement to their HRQoL than responders to treatment. Thus, restoring and/or maintaining quality of life should be an important goal of treatment.

HRQoL can be analyzed by universal or disease specific scales, the latter usually have better reactivity. Medical Outcomes Study Short Form 36 Health Survey (SF-36) is one of the most widely used universal HRQoL scales, and it is widely used in the HRQoL measurement of general population, evaluation of clinical trials and health policy evaluation. The ITP Participants Assessment Questionnaire (ITP-PAQ) was developed to assess disease-specific quality of life (QoL) in adults with ITP. It is a 44-item questionnaire that includes scales for physical health (symptoms, fatigue/sleep, bother, and activity), emotional health (psychological and fear), overall QoL, social activity, women's reproductive health, and work. The reliability and validity of these scales have been confirmed by a number of studies at home and abroad.

Therefore, the investigators conducted a real-world multicenter study using SF-36 and ITP-PAQ questionnaires to assess the HRQoL in participants with ITP in the real world, and analyze the influencing factors of HRQoL so as to provide a sufficient basis for clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. aged of 14-80 years.
3. Need or do not need treatments.

Exclusion Criteria:

1. Patients have any concomitant disease that could impact their quality of life significantly such as mental disorders
2. Severe medical condition (lung, hepatic or renal disorder) other than ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
3. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
4. Patients who are deemed unsuitable for the study by the investigator.

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 2016 to December 2018, ITP patients aged above 14 years will be enrolled in this study. They will be recruited in ten hospitals of Shandong province, China. Patients were eligible if they can finish the questionares correctly by themselves. Patients were excluded if they have any concomitant disease that could impact their quality of life significantly.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
ITP-PAQ | From date of randomization until the date of first documented progression,up to 12 months
  ITP Patient Assessment Questionnaire (ITP-PAQ) was developed to assess disease-specific quality of life (QoL) in adults with ITP. It is a 44-item questionnaire that includes scales for physical health (symptoms, fatigue/sleep, bother, and activity), emotional health (psychological and fear), overall QoL, social activity, women's reproductive health, and work.
SF-36 | From date of randomization until the date of first documented progression,up to 12 months
  Medical Outcomes Study Short Form 36 Health Survey (SF-36) is one of the most widely used universal HRQoL scales, and it is widely used in the HRQoL measurement of general population, evaluation of clinical trials and health policy evaluation.

SECONDARY OUTCOMES:
bleeding score | From date of randomization until the date of first documented progression,up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Shandong University Qilu hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambert MP, Gernsheimer TB. Clinical updates in adult immune thrombocytopenia. Blood. 2017 May 25;129(21):2829-2835. doi: 10.1182/blood-2017-03-754119. Epub 2017 Apr 17. PMID 28416506
- [Background] Grace RF, Neunert C. Second-line therapies in immune thrombocytopenia. Hematology Am Soc Hematol Educ Program. 2016 Dec 2;2016(1):698-706. doi: 10.1182/asheducation-2016.1.698. PMID 27913549
- [Background] Flores A, Klaassen RJ, Buchanan GR, Neunert CE. Patterns and influences in health-related quality of life in children with immune thrombocytopenia: A study from the Dallas ITP Cohort. Pediatr Blood Cancer. 2017 Aug;64(8). doi: 10.1002/pbc.26405. Epub 2017 Jan 23. PMID 28111877
- [Background] Efficace F, Mandelli F, Fazi P, Santoro C, Gaidano G, Cottone F, Borchiellini A, Carpenedo M, Simula MP, Di Giacomo V, Bergamaschi M, Vincelli ID, Rodeghiero F, Ruggeri M, Scaramucci L, Rambaldi A, Cascavilla N, Forghieri F, Petrungaro A, Ditonno P, Caocci G, Cirrincione S, Mazzucconi MG. Health-related quality of life and burden of fatigue in patients with primary immune thrombocytopenia by phase of disease. Am J Hematol. 2016 Oct;91(10):995-1001. doi: 10.1002/ajh.24463. Epub 2016 Jul 14. PMID 27351715
- [Background] Mathias SD, Li X, Eisen M, Carpenter N, Crosby RD, Blanchette VS. A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Effect of Romiplostim on Health-Related Quality of Life in Children with Primary Immune Thrombocytopenia and Associated Burden in Their Parents. Pediatr Blood Cancer. 2016 Jul;63(7):1232-7. doi: 10.1002/pbc.25984. Epub 2016 Apr 1. PMID 27037553